CLINICAL TRIAL: NCT03463252
Title: Value of Levonorgestrel-Releasing Intrauterine System (LNG-IUS) in the Fertility-preserving Treatment of Atypical Endometrial Hyperplasia and Early Endometrial Carcinoma
Brief Title: Value of LNG-IUS as Fertility-preserving Treatment of EAH and EC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Zheng Ying, Professor/Associate Director/Supervisor of Master Student, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHENG Ying
Record Dates: First submitted 2018-03-04; First posted 2018-03-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Cancer; Atypical Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia | interventions — Progesterone; Medroxyprogesterone Acetate; Gonadotropin-Releasing Hormone; ricin A-GnRH conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MPA for EC without progesterone contraindication (Active Comparator): The enrolled patient (endometrial cancer without contraindication of oral high dose progesterone) is allocated to one of three groups, MPA only, MPA+LNG-IUS, LNG-IUS only, by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if endometrial cancer is still present after 3 cycles.
  Interventions: Drug: Progesterone
- MPA+Mirena® for EC without contraindication (Experimental): The enrolled patient (endometrial cancer without contraindication of oral high dose progesterone) is allocated to one of three groups, MPA only, MPA+LNG-IUS, LNG-IUS only, by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if endometrial cancer is still present after 3 cycles.
  Interventions: Drug: Progesterone; Device: Mirena®
- Mirena® for EC without contraindication (Experimental): The enrolled patient (endometrial cancer without contraindication of oral high dose progesterone) is allocated to one of three groups, MPA only, MPA+LNG-IUS, LNG-IUS only, by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if endometrial cancer is still present after 3 cycles.
  Interventions: Device: Mirena®
- GnRH agonist+Mirena® for EC with contraindication (Active Comparator): The enrolled patient (endometrial cancer with contraindication of oral high dose progesterone) is allocated to either GnRH-a+ LNG-IUS or only LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if endometrial cancer is still present after 3 cycles.
  Interventions: Device: Mirena®; Drug: GnRH agonist
- Mirena® for EC with contraindication (Experimental): The enrolled patient (endometrial cancer with contraindication of oral high dose progesterone) is allocated to either GnRH-a+ LNG-IUS or only LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if endometrial cancer is still present after 3 cycles.
  Interventions: Device: Mirena®
- Mirena® for EAH without progesterone contraindication (Active Comparator): The enrolled patient (atypical endometrial hyperplasia without contraindication of oral high dose progesterone) is allocated to either MPA or LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if EAH is still present after 3 cycles.
  Interventions: Device: Mirena®
- MPA for EAH without progesterone contraindication (Experimental): The enrolled patient (atypical endometrial hyperplasia without contraindication of oral high dose progesterone) is allocated to either MPA or LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if EAH is still present after 3 cycles.
  Interventions: Drug: Progesterone
- Mirena® for EAH with progesterone contraindication (Active Comparator): The enrolled patient (atypical endometrial hyperplasia with contraindication of oral high dose progesterone) is allocated to either GnRH-a+ LNG-IUS or only LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if EAH is still present after 3 cycles.
  Interventions: Device: Mirena®
- GnRH-a+Mirena® for EAH with progesterone contraindication (Experimental): The enrolled patient (atypical endometrial hyperplasia with contraindication of oral high dose progesterone) is allocated to either GnRH-a+ LNG-IUS or only LNG-IUS by randomization. Continuous treatment for 3 months is one cycle. Hysteroscopic evaluation and biopsy will procedure every cycle. Patients with partial response or in stable condition, after 2 cycles, will receive continuous treatment for one more cycle again. Patients with complete response after 2 or 3 cycles are encouraged to pregnancy. The consideration of giving up fertility-sparing treatment is recommended: 1) if patient have documented progression on the biopsies; 2) if EAH is still present after 3 cycles.
  Interventions: Device: Mirena®; Drug: GnRH agonist

INTERVENTIONS:
Drug: Progesterone — MPA oral 250mg-500mg qd for 3 months per cycle
  Other Names: medroxyprogesterone acetate (MPA)
  Arms: MPA for EAH without progesterone contraindication; MPA for EC without progesterone contraindication; MPA+Mirena® for EC without contraindication
Device: Mirena® — levonorgestrel intrauterine sustained release system (LNG-IUS) placed in uterus for 3 months per cycle
  Other Names: LNG-IUS
  Arms: GnRH agonist+Mirena® for EC with contraindication; GnRH-a+Mirena® for EAH with progesterone contraindication; MPA+Mirena® for EC without contraindication; Mirena® for EAH with progesterone contraindication; Mirena® for EAH without progesterone contraindication; Mirena® for EC with contraindication; Mirena® for EC without contraindication
Drug: GnRH agonist — GnRH-a intramuscular injection 3.75mg once a month for 3 months per cycle
  Other Names: GnRH-a
  Arms: GnRH agonist+Mirena® for EC with contraindication; GnRH-a+Mirena® for EAH with progesterone contraindication

SUMMARY:
Primary end points:

This clinical trial is aimed to analyze the effectiveness of Levonorgestrel-Releasing Intrauterine System (LNG-IUS, Mirena®) in the fertility-sparing treatment of atypical endometrial hyperplasia and early endometrial carcinoma, including pathology response and pregnancy outcome.

Second end points:

To analyze the appearances of side-effects.

ELIGIBILITY:
For Patients With Endometrial Cancer：

Inclusion Criteria:

* ≤40 years of age:
* Having a strong desire for fertility preservation;
* Histological diagnosis is confirmed as well-differentiated (grade 1) endometrioid adenocarcinoma by the designated gynecological pathologists, and the progesterone receptors (PgRs) is positive in immunohistochemistry;
* Disease limited to the endometrium (stage 1A) on MRI;
* Serum CA125/199 level is within normal limit (Laparoscopic exploration to rule out ovarian tumor or another metastasis if necessary);
* Patients should have undergone counseling to learn fertility-preserving treatment is not standard of care for the treatment of EC, volunteered to participate in this study, signed the informed consent form, and agreed to participated in clinical follow-up.

Exclusion Criteria:

* Patients have allergies or contraindications (except for thromboembolic disease, liver dysfunction, hypertension, and diabetes) for the involved drugs;
* Patients have lynch syndrome (LS);
* Patients have contraindications for pregnancy;
* Patients have serious underlying disease, malignancies at other site(s), acute liver or kidney disease, acute liver or kidney diseases, acute or subacute genital tract infections and congenital or acquired abnormal uterine development (that may make intrauterine device placement impossible);
* Patients refuse to participate in clinical follow-up or sign the informed consent form.

For Patients With Endometrial atypical hyperplasia：

Inclusion Criteria:

* ≤ 40 years of age
* Having a strong desire for fertility preservation
* Histological diagnosis is confirmed as atypical endometrial hyperplasia (EAH) by the designated gynecological pathologists
* Having volunteered to participate in this study, signed the informed consent form, and agreed to participate in clinical follow-up

Exclusion Criteria:

* Patients have allergies or contraindications (except for thromboembolic disease, liver dysfunction, hypertension, and diabetes) for the involved drugs
* Patients have contraindications for pregnancy
* Patients have serious underlying disease, malignancies at other site(s), acute liver or kidney disease, acute or subacute genital tract infections, and congenital or acquired abnormal uterine development (that may make intrauterine device placement impossible)
* Patients refuse to participate in clinical follow-up or sign the informed consent form.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Response | 6-12 months
  Pathologic response to medicine treatment is categorized as complete response (CR), partial response (PR), no change (NC), and progressive disease (PD). CR is defined as the absence of any hyperplastic or cancerous lesion. PR is defined as the residual lesion with degeneration and atrophy of endometrial glands. NC is defined as residual lesion without degeneration or atrophy of endometrial glands. PD is defined as the appearance of endometrial cancer for EAH and grade 2 (G2) or 3 for EC.
Pregnancy Rate | 7-144 months
  The percentage of successful pregnancies in the CR patients.
Live Birth Rate | 16-144 months
  The percentage of successfully alive baby delivery in the pregnant patients.

SECONDARY OUTCOMES:
Side-Affects Rate | 1-144 months
  The appearances of side-effects include weight gain, irregular vaginal bleeding, breast pain, appetite changes, nausea, vomiting, rash, jaundice, thromboembolism, hypertension, liver dysfunction, kidney dysfunction, glucose intolerance, and diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ushijima K, Yahata H, Yoshikawa H, Konishi I, Yasugi T, Saito T, Nakanishi T, Sasaki H, Saji F, Iwasaka T, Hatae M, Kodama S, Saito T, Terakawa N, Yaegashi N, Hiura M, Sakamoto A, Tsuda H, Fukunaga M, Kamura T. Multicenter phase II study of fertility-sparing treatment with medroxyprogesterone acetate for endometrial carcinoma and atypical hyperplasia in young women. J Clin Oncol. 2007 Jul 1;25(19):2798-803. doi: 10.1200/JCO.2006.08.8344. PMID 17602085
- [Background] Rodolakis A, Biliatis I, Morice P, Reed N, Mangler M, Kesic V, Denschlag D. European Society of Gynecological Oncology Task Force for Fertility Preservation: Clinical Recommendations for Fertility-Sparing Management in Young Endometrial Cancer Patients. Int J Gynecol Cancer. 2015 Sep;25(7):1258-65. doi: 10.1097/IGC.0000000000000493. PMID 26186070
- [Background] Minig L, Franchi D, Boveri S, Casadio C, Bocciolone L, Sideri M. Progestin intrauterine device and GnRH analogue for uterus-sparing treatment of endometrial precancers and well-differentiated early endometrial carcinoma in young women. Ann Oncol. 2011 Mar;22(3):643-649. doi: 10.1093/annonc/mdq463. Epub 2010 Sep 28. PMID 20876910
- [Background] KELLEY RM, BAKER WH. Progestational agents in the treatment of carcinoma of the endometrium. N Engl J Med. 1961 Feb 2;264:216-22. doi: 10.1056/NEJM196102022640503. No abstract available. PMID 13752346
- [Background] Zhang Q, Qi G, Kanis MJ, Dong R, Cui B, Yang X, Kong B. Comparison among fertility-sparing therapies for well differentiated early-stage endometrial carcinoma and complex atypical hyperplasia. Oncotarget. 2017 May 3;8(34):57642-57653. doi: 10.18632/oncotarget.17588. eCollection 2017 Aug 22. PMID 28915701
- [Background] Wildemeersch D, Andrade A, Goldstuck N. Femilis((R)) 60 Levonorgestrel-Releasing Intrauterine System-A Review of 10 Years of Clinical Experience. Clin Med Insights Reprod Health. 2016 Aug 9;10:19-27. doi: 10.4137/CMRH.S40087. eCollection 2016. PMID 27547046
- [Background] Karimi-Zarchi M, Dehghani-Firoozabadi R, Tabatabaie A, Dehghani-Firoozabadi Z, Teimoori S, Chiti Z, Miratashi-Yazdi A, Dehghani A. A comparison of the effect of levonorgestrel IUD with oral medroxyprogesterone acetate on abnormal uterine bleeding with simple endometrial hyperplasia and fertility preservation. Clin Exp Obstet Gynecol. 2013;40(3):421-4. PMID 24283179
- [Background] Gallos ID, Shehmar M, Thangaratinam S, Papapostolou TK, Coomarasamy A, Gupta JK. Oral progestogens vs levonorgestrel-releasing intrauterine system for endometrial hyperplasia: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Dec;203(6):547.e1-10. doi: 10.1016/j.ajog.2010.07.037. PMID 20934679
- [Background] Orbo A, Vereide A, Arnes M, Pettersen I, Straume B. Levonorgestrel-impregnated intrauterine device as treatment for endometrial hyperplasia: a national multicentre randomised trial. BJOG. 2014 Mar;121(4):477-86. doi: 10.1111/1471-0528.12499. Epub 2013 Nov 28. PMID 24286192
- [Background] Kim MK, Seong SJ, Kim JW, Jeon S, Choi HS, Lee IH, Lee JH, Ju W, Song ES, Park H, Ryu HS, Lee C, Kang SB. Management of Endometrial Hyperplasia With a Levonorgestrel-Releasing Intrauterine System: A Korean Gynecologic-Oncology Group Study. Int J Gynecol Cancer. 2016 May;26(4):711-5. doi: 10.1097/IGC.0000000000000669. PMID 26905333
- [Background] Practice Bulletin No. 149: Endometrial cancer. Obstet Gynecol. 2015 Apr;125(4):1006-1026. doi: 10.1097/01.AOG.0000462977.61229.de. No abstract available. PMID 25798986
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO consensus conference on endometrial cancer: Diagnosis, treatment and follow-up. Radiother Oncol. 2015 Dec;117(3):559-81. doi: 10.1016/j.radonc.2015.11.013. Epub 2015 Dec 9. PMID 26683800
- [Background] Lee SW, Lee TS, Hong DG, No JH, Park DC, Bae JM, Seong SJ, Shin SJ, Ju W, Lee KH, Lee YK, Cho H, Lee C, Paek J, Kim HJ, Lee JW, Kim JW, Bae DS. Practice guidelines for management of uterine corpus cancer in Korea: a Korean Society of Gynecologic Oncology Consensus Statement. J Gynecol Oncol. 2017 Jan;28(1):e12. doi: 10.3802/jgo.2017.28.e12. Epub 2016 Oct 27. PMID 27894165
- [Background] Denny L, Quinn M. FIGO Cancer Report 2015. Int J Gynaecol Obstet. 2015 Oct;131 Suppl 2:S75. doi: 10.1016/j.ijgo.2015.06.024. No abstract available. PMID 26433677
- [Background] The American College of Obstetricians and Gynecologists Committee Opinion no. 631. Endometrial intraepithelial neoplasia. Obstet Gynecol. 2015 May;125(5):1272-1278. doi: 10.1097/01.AOG.0000465189.50026.20. PMID 25932867
- [Background] Chinese Medical Association Department of Gynecologic Oncology., Guidelines on Clinical Fertility-Sparing Treatment of Gynecologic Cancer. Chinese Journal of OBsterics and Gynecology, 2014(4):9-9
- [Background] NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®). Uterine Neoplasms. Version 2.2017 - April 25, 2017. NCCN.org
- [Background] Guidelines on Clinical Management of Endometrial Hyperplasia. HKCOG GUIDELINES NUMBER 631 (May 2015)
- [Background] Reproductive endocrinology group of China Health Industry Management Association for maternal and child health industry branch. consensus conference on endometrial hyperplasia: Diagnosis, treatment and follow-up. Journal of Reproductive Medicine. 2017. 26(10): p. 957-959.
- [Background] Ebina Y, Katabuchi H, Mikami M, Nagase S, Yaegashi N, Udagawa Y, Kato H, Kubushiro K, Takamatsu K, Ino K, Yoshikawa H. Japan Society of Gynecologic Oncology guidelines 2013 for the treatment of uterine body neoplasms. Int J Clin Oncol. 2016 Jun;21(3):419-34. doi: 10.1007/s10147-016-0981-1. Epub 2016 Apr 26. PMID 27116188
- [Background] Royal College of Obstetricians and Gynaecologists (RCOG) with the British Society for Gynaecological Endoscopy (BSGE). Management of Endometrial Hyperplasia. Green-top Guideline No. 67. RCOG/BSGE Joint Guideline. London; 2016 (cited 29 March 2016).
- [Derived] Mittermeier T, Farrant C, Wise MR. Levonorgestrel-releasing intrauterine system for endometrial hyperplasia. Cochrane Database Syst Rev. 2020 Sep 6;9(9):CD012658. doi: 10.1002/14651858.CD012658.pub2. PMID 32909630

DOCUMENTS (1):
  • Informed Consent Form (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03463252/ICF_000.pdf